CLINICAL TRIAL: NCT01999478
Title: Novel Biophotonics Methodology for Colon Cancer Screening
Acronym: BRP
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Hemant Kumar Roy, BMC Attending Physician, Boston Medical Center
Other Study IDs: R01CA128641 (NIH)
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing colonoscopy: Patients undergoing colonoscopy per standard of care.

SUMMARY:
The study is testing a new, safe and effective way for the early detection of colon cancer. The method uses Low-coherence Enhanced Backscattering Spectroscopy (LEBS). This is an optic probe which is a small device that uses light (not laser) to assess the colon lining. This probe will be used before colonoscopy to identify subjects who do and do not have precancerous changes in the colon by capturing the light reflected back from the rectal wall and that will be assessed without the need for colonoscopy and bowel preparation (colon cleaning). This device may detect early cancerous changes in colon tissue with higher accuracy than current tests.

DETAILED DESCRIPTION:
Supported by multiple grans from the NIH, we have developed and performed preliminarily clinical studies on a suite of biophotonics techniques that promises to have unprecedented accuracy in risk- stratification of colonic neoplasia. The main goal for this study is to establish a Bioengineering Research Partnership (BRP) with the objective to refine and provide comprehensive, definitive multi-center validation of these novel methodologies for colorectal cancer (CRC) screening, thus providing a quantum leap in population screening.

Colonoscopy has the potential of reducing colorectal cancer (CRC) occurrence by ~90% through the identification and interdiction of the precursor lesion, the adenomatous polyp. However, CRC remains the second leading cause of cancer deaths in the United States with an anticipated 153,760 new cases in 2007. The major reason why existing CRC screening strategy is not adequate is as follows:

According to existing recommendations, every patient over the age of 50 is considered at risk for CRC and is a candidate for colonoscopic surveillance to be performed at least every 10 years. However, screening the entire eligible population (>80 million Americans over age 50) through colonoscopy is practically impossible for a variety of reasons including expense (the financial burden on the health care would be ~$100B a year), patient reluctance, complication rate, and insufficient number of endoscopists. Indeed, currently only less than 20% of the population undergo colonoscopy. The potential solution to this could be risk-stratification. The lifetime incidence of colon polyps is ~20-30% and CRC is ~6%. Thus, instead of performing colonoscopy on the entire population, targeting the group at risk for developing neoplasia would allow the focusing of this finite endoscopic resource on subjects who will actually benefit from this invasive test. Current approaches at risk-stratification (e.g. flexible sigmoidoscopy, fecal occult blood test) are plagued by unacceptably poor sensitivity and positive predictive value. Thus, more accurate approaches are urgently needed to triage patients for colonoscopy. This test has to be considerably less expensive than colonoscopy (a colonoscopy costs ~$1,000-2,000), minimally invasive and performed by a primary care physician. (The strategy is analogous to the Pap-smear screening for cervical cancer: 50 years ago, cervical cancer used to be the first major cause of cancer deaths in women. The incidence was reduced by more than 70%, from number 1 killer in women to number 13, by introduction of the Pap-smear as an initial screening test. Currently, no such initial screening test is available in case of CRC.)

The proposed program is based on novel spectroscopic techniques developed by our multidisciplinary team, comprised of biomedical and electrical engineers, gastroenterologists, cancer biologists, and biostatisticians. Two techniques have been developed: low-coherence enhanced backscattering (LEBS) spectroscopy and four-dimensional elastic light scattering fingerprinting (ELF). Many screening techniques (e.g., flexible sigmoidoscopy) exploit the "field effect" of colon carcinogenesis, the proposition that the genetic/environmental milieu that results in a neoplastic lesion in one area of the colon should be detectable in uninvolved (i.e., colonoscopically normal-appearing) mucosa throughout the colon. Several lines of evidence suggest that nano/micro-architectural alterations are among the earliest pre-neoplastic markers of colon carcinogenesis.

Our group was the first to explore the concept of the field effect for cancer screening by means of optical examination of colonoscopically and histologically normal rectal tissue. A key capability of ELF and LEBS is that they sense these changes in microscopically normal tissue at a distance from a precancerous lesion. This opens up a possibility to identifying patients harboring adenomas in the colon by assessment of histologically and colonoscopically normal-appearing rectal mucosa without the need for colonoscopy.

We have completed successful animal and human studies showing that ELF and LEBS markers have superior performance to any existing markers of the field-effect of CRC. We have published the first demonstration that marked ELF/LEBS aberrations could be detected far earlier than any currently known markers of CRC including morphological (e.g. aberrant crypt foci, adenomas) or cellular (apoptosis, proliferation) markers. In our human studies, we demonstrated that the assessment of ELF/LEBS signatures in the endoscopically normal rectal mucosa (the most readily accessible colonic mucosa) accurately identified patients harboring neoplasia elsewhere in the colon. Indeed, the sensitivity of rectal ELF/LEBS was 100% for identifying the presence of adenomas elsewhere in the colon, far exceeding any previously described markers. This suggests that ELF/EBS could be exploited for CRC screening by means of a simple and inexpensive optical test without the need for either colonoscopy or bowel preparation.

Based on our preliminary data, we hypothesize that ELF/LEBS will be able to identify subjects who do and do not harbor adenomas in the colon based on optical alterations in the rectal mucosa that will be assessed without the need for colonoscopy and bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have appointments in the GI Clinic and are/or will be scheduled for an colonoscopy as per standard of care.
* Patients must be 18 years of age or older.

Exclusion Criteria:

* Patients who have a history of Inflammatory Bowel Disease.
* Patients who have colitis.
* Patients who are undergoing chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be obtained in the gastroenterology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2008-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Early cancer changes in the colon | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Vadim Backman, PhD, Principal Investigator — Northwestern University; Hemant Roy, MD, Principal Investigator — Boston University
Locations (5):
- United States (5):
  - University of Southern California, Los Angeles, California
  - NorthShore University HealthSystem, Evanston, Illinois
  - Northwestern Univeristy, Evanston, Illinois
  - University of Indiana, Indianapolis, Indiana
  - Boston Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No